CLINICAL TRIAL: NCT03963128
Title: Effectiveness of Vitamin D Supplementation to Reduce Injury and Illness in the UK Armed Forces With Specific Reference to Stress Fracture Risk Reduction
Brief Title: Vitamin D Supplementation in the Armed Forces
Acronym: D_SAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Surrey (Other)
Collaborators: Institute of Naval Medicine (Unknown); CTRM Lympstone (Unknown); Navy Command Headquarters (Unknown)
Responsible Party: Principal Investigator, Susan Lanham-New, Professor of Human Nutrition & Head, Nutritional Sciences Department, University of Surrey
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: D_SAF
Record Dates: First submitted 2019-05-17; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Stress Fracture; Injury
Keywords: Vitamin D; Royal Marines; Military Training; Illness
MeSH Terms: conditions — Fractures, Stress; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Recruited cohort divided into two groups: (i) a vitamin-D3 supplementation (50,000 IU administred every two months); and (ii) a placebo supplementation (administered orally every two months) control group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemented Vitamin D3 (Active Comparator)
  Interventions: Dietary Supplement: Supplementation Vitamin D3
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplementation Vitamin D3 — Supplementation of vitamin D3 at a dose of 50.000 IU administered every two months (equivalent of 800 IU per day)
  Arms: Supplemented Vitamin D3
Dietary Supplement: Placebo — Placebo administred every two months
  Arms: Placebo

SUMMARY:
The study will comprise of an original investigation that will take the form of a prospective intervention (two matched groups) study. Condition-1 will be a vitamin D supplementation group (50.000 IU every two months), and Condition-2 will be a placebo supplementation group.

The primary research aim of this project is to evaluate the effectiveness of vitamin D supplementation to reduce stress fracture risk and susceptibility to skin, soft tissue infection (SSTI) and respiratory infection in Royal Marine recruits undertaking arduous physical training in a randomised control trial (RCT). The secondary research aims are:

1. To investigate whether supplementation of vitamin D3 at a dose of 50.000 IU every two months (equivalent to 800 IU per day) is effective in reducing the risk of stress fracture and susceptibility to skin, soft tissue and respiratory infection.
2. To examine changes in vitamin D status (relative to baseline serum 25(OH)D concentration), serum PTH concentration, and markers of bone turnover in response to vitamin D3 supplementation during the winter and summer months.
3. To identify interactions between dietary intakes, physical fitness, physical characteristics (body mass, BMI, thigh girth), smoking habit, alcohol consumption, and stress fracture prevalence with serum 25(OH)D status, serum PTH concentration and markers of bone turnover in the vitamin D3 supplemented group vs. the placebo supplemented group.

DETAILED DESCRIPTION:
Study Overview:

Aim: The effect of vitamin D3 supplementation in (male) Royal Marine recruits during 32-weeks of (arduous) initial military training on stress fracture and respiratory illness risk. Volunteer recruits will initially complete a healthy history, smoking habit and alcohol consumption questionnaire. Height, body mass (from which BMI will be calculated), and calf girth/skinfold will be measured. A 20 ml blood sample will be drawn (gold and purple top vacutainers) for determination of vitamin D status, calcium and albumin concentrations, PTH concentration, markers of bone turnover, antibody responses against S. aureus or other antigens and plasma cytokine levels. A (3-5 ml) saliva sample will be taken for S. aureus culture, and for assessment of oral microbiota, cytokine and antibody levels in saliva. A dry swab would be taken from both anterior nares for enumeration of S. aureus, and stored in phosphate buffered saline. The study recruit cohort will be divided into two groups: (i) a vitamin-D3 supplementation (50,000 IU administered orally every two months - equivalent to 800 IU per day); and (ii) a placebo supplementation (administered orally every two months) control group. The vitamin D supplement and the placebo supplement will be manufactured by Pharmaterials Ltd., Unit B, 5 Boulton Road, Reading, RG2 0NH, UK. The active and placebo supplements will be presented as identical (size and appearance) tablets, indiscernible from each other for the volunteer or the study team in situ at CTC. Both groups will receive one tablet at each time point. Recruits will be randomly assigned to a study group, but the two groups will be matched for age, height, body mass and aerobic fitness. The randomisation of supplement/placebo administration to study volunteers will be undertaken by statisticians from the University of Surrey. Study team staff will monitor supplement taking and will further confirm supplement taking through exit interviews. Further 20 ml blood samples will be drawn every two months (i.e. at weeks 8, 16 and 32 of RM training), saliva samples and nasal swabs will also be taken, and the smoking habit and alcohol consumption questionnaire will be re-administered. The study team will take into consideration prevailing data on recruit attrition to inform this decision. Food Frequency Questionnaire (FFQ) will be administered in week-6 of training; this will allow the recruits' habitual RM training diet to be established following the civilian to military transition. Permission will be sought to collate the outcome of the week-1 and week-9 Royal Marine Fitness Assessment (RMFA). Permission will also be sought to prospectively collate data from the Defence Medical Information Capability Programme (DMICP) system describing the prevalence of injury and illness in study volunteers.

Study Procedures: All potential volunteer recruits to the study will have been initially passed medically and physically fit to undertake RM training. Following an initial brief, those recruits volitionally consenting to participate in the study will complete a Health History Questionnaire and a Smoking Habit and Alcohol Consumption Questionnaire. The Royal Marine Fitness Assessment (RMFA) is completed as part of the Recruit Syllabus (RS10) in weeks 1 and 9 of training; these data (i.e. Multi-Stage Fitness Test performance, number of sit-ups, number of press-ups and number of pull-ups) are collected by the PT Branch at CTC, and will be compiled by the study team to allow fitness comparisons to be made with the recruit sample monitored during SGBHP. Height and body mass will be measured (from which BMI will be calculated), and calf girth/skinfold will be measured, the Smoking Habit and Alcohol Consumption Questionnaire completed, antibiotic exposure determined (i.e. antibiotics use not prescribed by the Medical Centre will be ascertained, where the antibiotics prescribed by Medical Centre will be collected from medical centre notes), occurrence of skin infections treated outside the CTCRM Medical Centre determined (where skin infections diagnosed by Medical Centre will be collected from medical centre notes), and a further blood sample will be drawn every two months during training (i.e. at weeks 8, 16) and at the End of training (week32). The precise timing of measurement sessions will be determined through discussions between the study team and the Commando Training Wing (CTW). All measures will be undertaken in appropriate venues at CTC, and will be accommodated in the recruits' programme where there would be minimum impact upon other training/personal administration activities.

Vitamin D or Placebo Supplement Administration: The INM study team staff will undertake vitamin D or placebo supplement administration during a programmed medical serial in the RM recruit programme. The study team will observe and monitor recruits taking the supplement or placebo tablet, and will further confirm supplement or placebo taking through exit interviews. The pattern of randomisation of the supplement(s) and placebo for the study will be determined and monitored independently by UoS study team members. There will be two study groups - a vitamin D supplement group and a placebo supplement group. The two groups will be matched for age, height, body mass and aerobic fitness. The study plan is to supplement at the Start of Training, and every two months thereafter (i.e. at weeks 8, 16 and 24 of RM training). Preliminary discussions with CTC indicate that - to schedule this within the RM training programme and therefore ensure minimum impact on RM recruit time - supplementation during training may need to take place at weeks 6, 15 and 24. During these programmed serials, the study team will also collate information detailing if a study participant had undertaken military exercises or leave, where they would be exposed to increased sunlight, since the last measurement time point. This will be particularly pertinent where measurement points span CTC block leave (i.e. Christmas, Easter and Summer).

Assessment of Injury/Illness Incidence: The incidence of injury/illness (including SF, SSTI and respiratory infection) in recruits during training will be monitored in association with colleagues from the Medical Centre.

Measurements:

1. Health History Questionnaire: Whilst attending for the blood sample, a Health History Questionnaire will be completed.
2. Smoking and Alcohol Histories Questionnaire: Whilst attending for the blood sample, a validated Smoking and Alcohol Histories Questionnaire will be completed.
3. Body Mass: Volunteers will be weighed in shorts and t-shirt to the nearest 0.1 kg (Seca, Hamburg, Germany).
4. Height: Volunteers will remove their shoes/boots before standing on the stadiometer (Invicta, England) with feet together. Feet, buttocks and scapulae will be in contact with the back of the stadiometer, and personnel should look directly ahead. Height will be measured to the nearest 0.1 cm.
5. Body Mass Index (BMI): Body mass index will be calculated according to the equation, BMI = Body Mass ÷ (Height)2.
6. Calf Circumference: Each recruit will be measured to the nearest 0.1 cm at the site of maximum girth using a Silverflex anatomical metal tape measure (Rabone Chesterman, England).
7. Calf Skinfold: A calf skinfold will be measured to the nearest 0.2 mm at the site of maximum girth for each recruit using Harpenden callipers (BodyCare UK).
8. Royal Marine Fitness Assessment (RMFA): The RMFA is a programmed serial of RM training, and is administered in weeks 1 and 9 of training. It comprises four component parts including: Multistage Fitness Test (MSFT); press-up test; sit-up test; and pull-up test. The RMFA will be administered by the PT Branch in accordance with CTC PT Instructional Specifications (ISPECs). The MSFT will be employed to estimate maximum oxygen uptake (VO2max). Sit-ups, press-ups, and pull-ups will be performed in accordance with standard RM techniques.
9. MOD Food Frequency Questionnaire (FFQ): A questionnaire examining nutrition and physical activity levels during the childhood and teenage years, and validated for use in military recruits, will be administered during a classroom serial in week-6 of training. This questionnaire was originally developed to assess nutritional and lifestyle influences on bone health in pre-menopausal women, and is based on a FFQ approach. Output data provide an estimated dietary analysis of respondents (in terms of macroand micro-nutrient intakes), and information on other lifestyle risk factors associated with bone health including physical activity habits and smoking. The aim of the FFQ is to classify research participants into low, medium and high consumers of dairy and vegetables. Non-dietary questions based on previous physical activity levels are calculated using James and Schofield equations. Questions regarding smoking are also included. In order to make this questionnaire more appropriate for the MOD population, certain regional food items were omitted, questions about convenience and takeaway food consumption were included, and questions regarding alcohol intake were modified to reflect the customary alcoholic beverages of the target age group in the present study (e.g. Alco-pops). The James and Schofield Human Energy Requirement equation will be used to calculate basal metabolic rate (BMR),31 from which the mean energy intake (EI) to BMR ratio (EI:BMR) will be determined to assess reporting accuracy of dietary intake. Goldberg et al.32 established a EI:BMR ratio of 1.35 as being indicative of food diary under-reporting.
10. Saliva: A (3-5 ml) saliva sample will be taken for S. aureus culture, and for assessment of oral microbiota, cytokine and antibody levels in saliva.
11. Nasal Swab: A dry swab will be taken from both anterior nares for enumeration of S.aureus, and stored in phosphate buffered saline.
12. Measures of metabolic and/or biochemical status: A 20 ml blood sample will be drawn from an antecubital vein by medical personnel - using gold and white capped vacutainers - during routine medical serials at the Start and End of Training, and during scheduled medical serials at weeks 8, 16 (or 6, 15) of training to match the weeks when the supplement/placebo will be administered. The 15 ml gold vacutainer blood samples will be left to clot for 1 h, after which it will be centrifuged for 15 min within 1 - 2 h, the serum subsequently being aspirated and initially stored in plastic 0.5 ml aliquots in plastic Eppendorf tubes at -80 C at CTC. The white vacutainer tubes contain EDTA, which acts as a strong anticoagulant for whole blood samples. The blood will be centrifuged for 15 min and the plasma supernatant will be extracted and initially stored in plastic 0.5 ml aliquots in plastic Eppendorf tubes at -80 C at CTC. The serum samples will be assayed for: vitamin D status (relative to 25(OH)D); parathyroid hormone (PTH) concentration; calcium (Ca) and albumin (as markers of vitamin D status and Ca metabolism); serum collagen type I cross-linked C-telopeptide (CTx) as a marker of bone resorption; carboxy-terminal propeptide of type I collagen (P1NP) as a marker of bone formation (as markers of bone turnover); and ferritin (Fe) as a marker of iron status. Immunological metrics will be measured in serum including: serum cytokine levels; antibody responses against S. aureus or other antigens; full blood count; lymphocyte phenotyping and measurement of T cell responses against S.aureus and S. pyogenes antigens; and RNA profiling. At one sample point only, specific DNA would be extracted from the cell pellet acquired from the (white top EDTA vacutainers) blood sample, which has been centrifuged to acquire plasma. This DNA will be analysed ONLY to study the genetic variation in the calcium / vitamin D axis in recruit volunteers. The specific SNPs for analysis will include: rs12785878 - 11q12 near DHCR7 (7-dehydrocholesterol reductase); rs10741657 - 11p15 near CYP2R1 (25hydroxylation); rs2282679 - 4p12 in GC (vitamin D binding protein); rs1998199 - 20q13 near STX16/NPEPL1/GNAS (associated with pseudo-hypoparathyoidism); rs6013897 - 20q13 near CYP24A1 (24 hydroxylation); and, Apa, taq, Bsm, fok1 - vitamin D receptor gene polymorphism. Samples for DNA extraction and analysis will initially be transferred to the University of Oxford, Oxford, for this work to be completed.
13. Microbiological assessment of aetiology: If a purulent discharge is evident, microbiological swabs will be obtained from infected lesions, swabs being either taken on the surface (where no incision and drainage occurs) or from pus samples (where Incision and drainage has occurred). These will be cultured for S. aureus as recommended in the current UK Standards in Microbiological Investigation. Consent for collection of any such samples from NHS laboratories to which they may have been sent will be obtained at baseline. Additionally, serological diagnosis will be determined using anti-S. aureus and anti-S. pyogenes antigen EIAs, including the methods described (Karppelin, 2015; Toleman, 2015; Jeng, 2010).
14. Incidence of illness and injury relative to week of training: The incidence of injury/illness (including SF, SSTI and respiratory infection) in recruits during training will be monitored in association with colleagues from the Medical Centre. Consent to prospectively access this medical information will be obtained from recruits at the start of training, and their consent will be re-confirmed at the end of training in the event of any circumstances having changed. Recruits participating in the study, who report to the Medical Centre, will have the details of their complaint coded on the DMICP system by the doctor, nurse or medical assistant according to current CTC procedures. In addition the staff member will categorise the presenting complaint as 'Injury' or 'Illness or Disease' according to the DMICP read codes. The Week of Training will also be coded on DMICP. To ensure data protection issues are addressed and to ensure recruit confidentiality, all medical data relating to illness/injury will be collated through a routine meeting with a single point of contact in the Medical Centre. The DMICP database will be searched for recruits participating in the study who have attended medical appointments; the categorisation of the presenting complaint and Week of Training will be identified. As this study is concerned with the recruit outcomes to training in itsentirety, recruits who enter Hunter Company due to the severity of their illness/injury - or for professional reasons - will continue to participate in the study (subject to their continued consent), and progress with their new Troop will be mapped through to passout. As far as possible SSTI will be systematically categorised as follows:

i. Impetigo: A skin infection that is common throughout the world, consists of discrete purulent lesions caused by beta haemolytic Streptococcus or S. aureus.

ii. Cutaneous Abscesses: Collections of pus within the dermis and deeper skin tissues.

iii. Furuncles and Carbuncles: Furuncles "boils" are infections of the hair follicles caused by S. aureus in which suppuration extends through the dermis into the subcutaneous tissue where a small abscess forms. A carbuncle is a collection of infected hair follicles and can occur anywhere on hairy skin.

iv. Folliculitis: Superficial inflammation and pus is present in the epidermis. v. Cellulitis and Erysipelas: Diffuse spreading skin infections excluding infections associated with underlying suppurative foci such as cutaneous abscesses, NF, septic arthritis and osteomyelitis. Erysipelas affects the upper dermis and cellulitis the deeper dermis and subcutaneous fat. Erysipelas and cellulitis are usually due to Streptococcus pyogenes.

vi. Necrotising SSTI: Rare subcutaneous infection that tracks along the fascial planes and may involve the muscle, fat and deeper structures, with an associated mortality of up to 83% if associated with toxic shock. The major pathogens are S. pyogenes and S. aureus.

vii. Other SSTI not classified.

ELIGIBILITY:
Inclusion Criteria:

* Royal Marines
* aged between 16 - 32 years at the Start of Training,
* successfully completed the physical and professional selection tests which comprise the Potential Royal Marine Course (PRMC), and be deemed medically fit and healthy following medical screening at the AFCO and again at CTC if required.

Exclusion Criteria:

* not participating in Recruit Syllabus (RS10) for RM recruit training
* deemed unsuitable by the IMO or the training team.

Ages: 16 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4450 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of supplementation of vitamin D3 at a dose of 50.000 IU administered every two months (equivalent of 800 IU per day) in reducing the risk of stress fracture. | 32 weeks

SECONDARY OUTCOMES:
The effectiveness of supplementation of vitamin D3 at a dose of 50.000 IU administered every two months (equivalent of 800 IU per day) in reducing the risk of susceptibility to skin infection. | 32 weeks
The effectiveness of supplementation of vitamin D3 at a dose of 50.000 IU administered every two months (equivalent of 800 IU per day) in reducing the risk of susceptibility to soft tissue (SSTI) infection. | 2018 - 2023
The effectiveness of supplementation of vitamin D3 at a dose of 50.000 IU administered every two months (equivalent of 800 IU per day) in reducing the risk of respiratory infection. | 32 weeks
Changes in vitamin D status (relative to baseline serum 25(OH)D concentration) in response to vitamin D3 supplementation during the winter and summer months. | 32 weeks
Changes in serum PTH concentration (relative to baseline concentration) in response to vitamin D3 supplementation during the winter and summer months. | 32 weeks
Changes in markers of bone turnover (relative to baseline concentration) in response to vitamin D3 supplementation during the winter and summer months. | 32 weeks
Interactions between dietary intakes, physical fitness, physical characteristics, smoking habit, alcohol consumption, and stress fracture prevalence with serum 25(OH)D status. | 32 weeks
Interactions between dietary intakes, physical fitness, physical characteristics, smoking habit, alcohol consumption, and stress fracture prevalence with serum PTH concentrations. | 32 weeks
Interactions between dietary intakes, physical fitness, physical characteristics, smoking habit, alcohol consumption, and stress fracture prevalence with markers of bone turnover. | 32 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Naval Medicine, Gosport, United Kingdom

IPD SHARING:
Plan to Share IPD: No